CLINICAL TRIAL: NCT00836043
Title: Safety, Effectiveness and Patient Acceptance of the Treatment With MabCampath in Chronic Lymphocytic Leukemia (CLL)
Brief Title: Safety, Effectiveness and Patient Acceptance of the Treatment With MabCampath in Chronic Lymphocytic Leukemia
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to low enrollment.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: 13418; 13858; 14241; MC0701; STAR
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; alemtuzumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Alemtuzumab (MabCampath)

INTERVENTIONS:
Drug: Alemtuzumab (MabCampath) — Intravenous therapy according to product information.
  Other Names: BAY86-5045

SUMMARY:
This study will collect data on safety, effectiveness and patient acceptance of MabCampath treatment under daily life conditions.

DETAILED DESCRIPTION:
As of 29 May 2009, the clinical trial sponsor is Genzyme Corporation. NOTE: This study was originally posted by sponsor Schering AG, Germany, which was subsequently renamed to Bayer Schering Pharma AG, Germany.

ELIGIBILITY:
Inclusion Criteria:

In- and outpatients suffering from CLL, who are treated with Mab Campath, and are routinely monitored with PCR (Polymerase Chain Reaction) for CMV infection during MabCampath treatment and for at least 2 months following completion of treatment.

Exclusion Criteria:

In accordance with Summaries of Product Characteristics (SPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients,who are suffering from chronic lymphocytic leukemia (CLL) and are treated with alemtuzumab (MabCampath)
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Efficacy related variables are patient's condition, physician's assessment of efficacy and tolerability, information whether application could be completed, clinical and laboratory findings. Safety Variables. | After first cycle of treatment, e.g. 12 weeks, then after 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- Many Locations, Bosnia and Herzegovina
- Many Locations, Israel
- Many Locations, North Macedonia